CLINICAL TRIAL: NCT06053060
Title: Evaluation of the Positioning of the Dynacup Cup "One C" Versus Standard Dynacup
Brief Title: Evaluation of the Positioning of the Dynacup Cup "One C" Versus "Standard Dynacup"
Acronym: DYNACUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, SMARMOR, MD, Groupe Hospitalier Diaconesses Croix Saint-Simon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ID RCB : 2020-A02843-36
Record Dates: First submitted 2023-03-24; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hip; Arthropathy
Keywords: One-C; Stadard; Dynacup
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Dynacup (Other): Hip arthroplasty with a standard Dynacup cup
  Interventions: Other: Randomisation Standard Dynacup or Dynacup One C
- Dynacup One C (Other): Hip arthroplasty with a cup Dynacup One C
  Interventions: Other: Randomisation Standard Dynacup or Dynacup One C

INTERVENTIONS:
Other: Randomisation Standard Dynacup or Dynacup One C — Randomisation

SUMMARY:
The ceramic-ceramic friction pair is widely used today in total hip arthroplasty, including fourth-generation ceramics which show the lowest wear rate. These have considerably reduced the risk of head fracture compared to previous generations; however, the risk of insert rupture persists with rates similar to those of third generation ceramics.

These ceramic fractures require complex revision surgery, which brings complications, exposing patients to the risk of third-body wear and tear related to persistent post-surgical debris. They are frequently due to an incorrect assembly of the ceramic causing intraoperative or early postoperative rupture. To fix this, manufacturers have developed pre-assembled cups in the factory. The Dynacup One C cup developed by Corin® corresponds to the pre-assembled version of the Dynacup cup, making it possible to eliminate the risk of anomaly during intraoperative assembly linked to the human factor and to offer patients with very small cups an adapted ceramic implant. A single study with a small sample compared the two implants (pre-assembled version [vs] modular version) clinically, radiologically and functionally without showing any significant difference. The lack of data in the literature comparing these two implants motivated us to conduct a randomized comparative study on a large sample of patients.

DETAILED DESCRIPTION:
Patients eligible for a total hip arthroplasty with a ceramic-ceramic friction couple and scheduled for surgery will be included in this study after information and collection of written consent.

After randomization, a preoperative radiograph with a calibration ball will be taken to plan the prosthesis and identify the characteristics of the operated hip.

An x-ray of the pelvis with a 28 mm ball will be carried out the day after the intervention according to the same preoperative procedures in order to measure the postoperative radiographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult man and woman > 18 years old
* Indication for hip arthroplasty with a Dynacup One C or standard Dynacup cup
* Patient informed of the study and signed a consent form

Exclusion Criteria:

* Refusal to participate in the study
* Indication of a friction couple other than ceramic-ceramic
* Contraindication or the technical impossibility of implanting an impacted acetabular component
* Pregnant or breastfeeding women.
* Minor patients aged < 18 years
* Subjects not affiliated to the national health insurance or to an equivalent insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
To Compare the positioning accuracy of the Dynacup One C (pre-assembled version) with that of the standard Dynacup. | Perioperative
  Radiographic measurement of the position of the center of rotation of the final implant, its inclination and its anteversion, compared to the positioning planned before the intervention for the 2 types of implants.

SECONDARY OUTCOMES:
To describe the rate of intraoperative secondary re-impactions of both groups | Perioperative
  Note the attempts at re-impactions for sensation of extrusion: after palpation with forceps of the bottom of the acetabulum (bone space - metal back for the standard Dynacups) or of its protruding periphery of the bone (for the pre-assembled versions) .
  ○ Note the operator's feeling before postoperative control X-ray on the good impaction of the acetabulum: at the bottom, doubtful or extrus.
To describe the rate of intraoperative complications according to the type of implant | Perioperative
  Describe the rate of intraoperative complications according to the type of implant:
  * Fracture of ceramics on impaction or assembly
  * Fracture of the bony acetabulum or unplanned acetabular protrusion
To describe the rate of insufficient impaction of the acetabulum in both groups | Perioperative
  Describe the rate of insufficient impaction of the acetabulum in the 2 versions
  * Radiographic measurement of the space between the bottom of the prosthetic acetabulum and the bottom of the milled bone acetabulum (Space > 2mm = impaction defect)
  * Radiographic analysis of postoperative front and side views by an independent evaluator
Indentify predictors for insufficient impaction of the acetabular implant | Perioperative
  Look for predictive factors of insufficient impaction of the acetabular implant
  * Depending on the type of implant
  * According to the morphology of the arthritic hip:
    * Type of indication and acetabular osteoarthritis: necrosis, upper lateral osteoarthritis, postero-internal osteoarthritis, global osteoarthritis or coxitis
    * Acetabular morphology: osteophytosis, dysplasia, osteocondensation, protrusion, sheathing
    * Femoral morphology: Dorr classification, cervico-diaphyseal angle.

CONTACTS AND LOCATIONS:
Overall Officials: Simon MARMOR, MD, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Dianconesses croix saint Simon, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No